CLINICAL TRIAL: NCT05660655
Title: Efficacy and Safety of Baricitinib in Different Doses for the Treatment of Moderate to Severe Rheumatoid Arthritis
Brief Title: Efficacy and Safety of Baricitinib for the Treatment of Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Md. Sadikul islam, Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU/2022/11646
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
Keywords: baricitinib; RA; JAKi
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Baricitinib 2mg and methotrexate 10mg (Active Comparator): Baricitinib 2mg once daily plus methotrexate 10mg per week
  Interventions: Drug: Baricitinib 2 MG
- Baricitinib 4mg and methotrexate 10mg (Experimental): Baricitinib 4mg once daily plus methotrexate 10mg per week
  Interventions: Drug: Baricitinib 4 MG Oral Tablet

INTERVENTIONS:
Drug: Baricitinib 4 MG Oral Tablet — baricitinib 4 mg once daily
  Other Names: for group B
  Arms: Baricitinib 4mg and methotrexate 10mg
Drug: Baricitinib 2 MG — baricitinib 4mg once daily in group A
  Other Names: for group A
  Arms: Baricitinib 2mg and methotrexate 10mg

SUMMARY:
This is a randomized controlled study. Baricitinib 4mg in one arm and Baricitinib 2mg in another arm will be used. Methotrexate 10mg per week in both arms will be used.

DETAILED DESCRIPTION:
This open label randomized controlled clinical trial will be conducted in the department of Rheumatology, BSMMU. The rheumatoid arthritis patients with moderate to severe disease activity (DAS 28 ESR/CRP>3.2) despite treatment with methotrexate or other csDMARDs will be considered as primary entry criteria for this study. Simple random sampling method will be applied. After a washout period of three weeks, Group A will be put on baricitinib 2 mg once daily and Group B will be put on baricitinib 4 mg once daily. Methotrexate 10mg will be used on both groups in addition to barcitinib. NSAIDs and adjuvant analgesics will be used if needed. All the patients will go through baseline evaluation before treatment which include-Disease Activity Score derivative for 28 joints (DAS 28ESR/CRP), Clinical Disease Activity Index (CDAI), Simplified Disease Activity Index (SDAI), Health Assessment Questionnaire-Disability Index (HAQ-DI) and laboratory tests like CBC, CRP, SGPT, Serum Creatinine, LDH, RF, ACPA, Chest X-ray P/A view and TST or interferon gamma release assay (IGRA). Follow up will be done at 4th, 12th and 24th week. Response to treatment will be evaluated by DAS 28 ESR/CRP. Primary endpoint for efficacy will be assessed at the end of 24th week by DAS 28 CRP response. Secondary endpoints will be determined by SDAI, CDAI and HAQ-DI. Adverse effects will be assessed by history, physical examinations and investigations

ELIGIBILITY:
Inclusion Criteria:

1. age greater than 18 years
2. patients fulfill the ACR/EULAR 2010 classification criteria for RA
3. DAS-28 CRP more than 3.2 despite optimum dose of methotrexate

Exclusion Criteria:

1. Recent or concurrent infection including active or latent tuberculosis except patients with latent tuberculosis in whom treatment was commenced ≥ 4 weeks before randomization
2. Hemoglobin (Hb) < 8 g/dl
3. White blood cell count < 4000, Neutrophil count < 1000, Platelet count < 100000/mm3
4. Live vaccines within 3 months prior to the first dose
5. Serum creatinine > upper limit of normal reference range
6. eGFR < 60 ml/minute/1.73 m2
7. Alanine transaminase (ALT) more than ULN
8. Pregnant or breast feeding females of child-bearing potential
9. Evidence or history of malignancy, with the exception of adequately treated or excised non-metastatic basal or squamous cell cancer of the skin or cervical carcinoma in situ
10. New York Heart Association Class III and IV congestive heart failure
11. Previous history of thromboembolism, deep venous thrombosis, diverticulitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Disease activity score 28-C-reactive protein (DAS28-CRP) | 6 months
  Disease activity score in 28 joints has to measure at 6 months. score less than or equal 3.2 will be regarded as low disease activity

SECONDARY OUTCOMES:
Clinical Disease activity index (CDAI) | 6 months
  clinical disease activity index at 6 months will be recorded. Score of equal or less than 10 will be regarded as low disease activity
Health Assessment Questionnaire-Disability Index (HAQ-DI) | 6 months
  health assesment by HAQ-DI at 6 months will be recorded. reduction of more than 0.22 will be regarded as improvement.
Disease activity score 28-C-reactive protein (DAS28-CRP) | 6 months
  Disease activity score in 28 joints has to measure at 6 months. score less than or equal 3.2 will be regarded as low disease activity

CONTACTS AND LOCATIONS:
Overall Officials: Sadikul i sadik, MBBS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Dr. Md. Sadikul islam, Dhaka, [Other], Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Genovese MC, Kremer JM, Kartman CE, Schlichting DE, Xie L, Carmack T, Pantojas C, Sanchez Burson J, Tony HP, Macias WL, Rooney TP, Smolen JS. Response to baricitinib based on prior biologic use in patients with refractory rheumatoid arthritis. Rheumatology (Oxford). 2018 May 1;57(5):900-908. doi: 10.1093/rheumatology/kex489. PMID 29415145
- [Result] Fleischmann R, Schiff M, van der Heijde D, Ramos-Remus C, Spindler A, Stanislav M, Zerbini CA, Gurbuz S, Dickson C, de Bono S, Schlichting D, Beattie S, Kuo WL, Rooney T, Macias W, Takeuchi T. Baricitinib, Methotrexate, or Combination in Patients With Rheumatoid Arthritis and No or Limited Prior Disease-Modifying Antirheumatic Drug Treatment. Arthritis Rheumatol. 2017 Mar;69(3):506-517. doi: 10.1002/art.39953. PMID 27723271
- [Result] Dougados M, van der Heijde D, Chen YC, Greenwald M, Drescher E, Liu J, Beattie S, Witt S, de la Torre I, Gaich C, Rooney T, Schlichting D, de Bono S, Emery P. Baricitinib in patients with inadequate response or intolerance to conventional synthetic DMARDs: results from the RA-BUILD study. Ann Rheum Dis. 2017 Jan;76(1):88-95. doi: 10.1136/annrheumdis-2016-210094. Epub 2016 Sep 29. PMID 27689735